CLINICAL TRIAL: NCT03690583
Title: Assessment of the Immunomodulatory Effect of Zinc Supplementation on the Clinical Evolution of Children With Pneumonia
Brief Title: Immunomodulation by Zinc Supplementation in Children With Pneumonia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universidad Nacional Autonoma de Mexico (Other)
Collaborators: Hospital General de Mexico (Other Government); Hospital Pediatrico de Coyoacan (Unknown)
Responsible Party: Principal Investigator, Rosa Maria Wong Chew, Professor B. Head of the Infectious Diseases Research Laboratory, Universidad Nacional Autonoma de Mexico
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CONACYT SALUD 2012-01-182274
Record Dates: First submitted 2018-09-20; First posted 2018-10-01 (Actual); Last update posted 2018-10-01 (Actual); Status verified 2018-09

CONDITIONS: Pneumonia; Children, Only
Keywords: Pneumonia; Zinc supplementation; Cytokines; Lymphoproliferation; Viruses; Respiratory bacteria
MeSH Terms: conditions — Pneumonia; Virus Diseases | interventions — Zinc Sulfate; Zinc; Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zinc group (Experimental): Zinc sulfate 10 mg in children younger than 1 year old, 20 mg in children older than 1 year old
  Interventions: Drug: Zinc sulfate
- Placebo group (Placebo Comparator): Glucose
  Interventions: Other: Glucose

INTERVENTIONS:
Drug: Zinc sulfate — Zinc sulfate 10 mg for children younger than 1 year old, 20 mg for children older than 1 year old, will be diluted in 1 ml of sterile water and administered orally every day in the morning during hospitalization
  Other Names: Zinc
  Arms: Zinc group
Other: Glucose — The placebo group will receive glucose diluted in 1 ml of sterile water orally every day during hospitalization
  Arms: Placebo group

SUMMARY:
Pneumonia is one of the main causes of morbidity and mortality in the world, especially in developing countries like ours.

The National Health and Nutrition Survey of Mexico, in 2006 showed underweight in 472,890 (5%) children under five years, low height in 1,194,805 (12.7%) and wasting in153,000 (1.6%) children. Zinc is decreased in malnutrition and is an essential cofactor for many proteins involved in cellular processes. Zinc deficiency leads to a decrease in the number of T cells, the ratio of Th1 to Th2 cells and the production of Th1 cytokines such as interferon gamma, with alteration in T cell mediated immunity. In malnourished children zinc supplementation restores the immune response. Reports of zinc supplementation in children with pneumonia are controversial.

The aims of this study are to evaluate the immunomodulatory effect of zinc supplementation in the clinical course of children with pneumonia, to evaluate the lymphoproliferative and cytokine response in these children and to explore whether the viral or bacterial etiology is related to the clinical response to supplementation with this micronutrient.

A clinical, randomized, prospective, controlled, double blinded study will be carried out. Children from 1 month to 5 years of age will be included, with the clinical and / or radiological diagnosis of pneumonia that enter the emergency room of the participant institutions. Empirical treatment for pneumonia will begin and each patient will be randomized 1:1 in 2 groups. One will receive zinc supplementation and another a placebo (glucose). Samples will be taken to determine the etiology (nasal lavage for multiplex polymerase chain reaction for 16 respiratory viruses and 6 bacteria) and a blood sample to measure the cytokine pattern and the lymphoproliferative response. After 7 days of treatment, a second sample will be taken for immunological studies (cytokine pattern and lymphoproliferative response). The following parameters will be measured to evaluate the clinical evolution: respiratory rate, temperature, oxygen saturation, inability to eat, duration of cough, rales, temperature normalization time, normalization time of oxygen saturation, normalization time of the respiratory rate, hospitalization time and outcome (discharge due to clinical improvement or death). A correlation will be made between the improvement in clinical parameters and mortality in the zinc supplementation group and the probable bacterial or viral etiology.

DETAILED DESCRIPTION:
Background: Pneumonia is one of the main causes of morbidity and mortality in the world, especially in developing countries like ours. Of an estimated 8.795 million deaths in children under 5 in the world in 2008, 68% were infectious causes, with the highest percentage due to pneumonia in 18%, followed by diarrhea in 15% and malaria in 8%, 41% of the deaths were in neonates, pneumonia being the 4th cause of death in this age group. Acute respiratory infections, diarrhea and malnutrition together cause 10% of deaths among children under 1 year of age. In Mexico, a pneumonia mortality rate of 120 per 100,000 inhabitants is reported in children under 1 year of age, and 5 deaths per 100,000 inhabitants in children from 1 to 4 years of age in 2007.

The results of the National Health and Nutrition Survey (ENSANUT), carried out in 2006 by the National Institute of Public Health, showed that 472,890 children under five years of age were classified as underweight (5%), 1,194,805 with low height (12.7%) and around 153,000 children with wasting (1.6%). The overall prevalence of anemia in urban areas was 22.8%, while in rural areas was 26.1%. Likewise, it is known that there are specific deficiencies of some micronutrients, such as vitamin A, C, E, zinc, iron, folic acid and iodine, among others. Malnourished children loose between 12 and 15% of their intellectual potential, have a higher risk of infectious diseases 8 to 12 times more than a healthy child and are more prone to chronic degenerative diseases. Malnutrition causes among others an effect of immunosuppression. One of the micronutrients that is decreased in malnutrition is zinc. Zinc is an essential cofactor for many proteins involved in cellular processes such as differentiation, proliferation and apoptosis. During zinc deficiency, the development of T lymphocytes, the polarization in effector cells and their function are altered. This leads to a decrease in the number of T cells, a decrease in the ratio of Th1 to Th2 cells with a decrease in the production of Th1 cytokines such as interferon gamma, and alteration in the defense mediated by T cells. In malnourished children zinc supplementation restores the immune response. Reports of zinc supplementation in children with infectious diseases are controversial. A study in Uganda reports that supplementation with zinc in children from 6 months to 5 years of age with severe pneumonia decreased the mortality from 12% to 4%, with a relative risk reduction of 0.67. Cellular immunity plays a very important role in the defense of the host against viruses and bacteria, zinc supplementation in children who have some degree of malnutrition and who suffer a serious infection could improve the immune response and improve the ability to respond to acute infection.

The aim of this study is to evaluate the immunomodulatory effect of zinc supplementation in the clinical course of children with pneumonia, to evaluate the lymphoproliferative and cytokine response in these children and to explore whether the viral or bacterial etiology is related to the clinical response to supplementation with this micronutrient.

Methods: This is a clinical, randomized, prospective, controlled, double blinded study. Children from 1 month to 5 years of age will be included, with the clinical and / or radiological diagnosis of pneumonia that enter the emergency room of the participant institutions. Empirical treatment for pneumonia will begin and each patient will be randomized 1:1 in 2 groups. One will receive zinc supplementation (10 mg of zinc sulfate in children younger than 1 year old and 20 mg of zinc sulfate in children older than 1 year old) and another a placebo (glucose 10 mg). Samples will be taken to determine the etiology (pharyngeal exudate, nasal lavage for multiplex polymerase chain reaction for 16 respiratory viruses and 6 bacteria) and a blood sample to measure the cytokine pattern and the lymphoproliferative response. After 7 days of treatment, a second sample will be taken for immunological studies (cytokine pattern and lymphoproliferative response). The following parameters will be measured to evaluate the clinical evolution: respiratory rate, temperature, oxygen saturation, inability to eat, duration of cough, crackling, temperature normalization time, normalization time of oxygen saturation, normalization time of the respiratory rate, hospitalization time and outcome (discharge due to clinical improvement or death). A correlation will be made between the improvement in clinical parameters and mortality in the zinc supplementation group and the probable bacterial or viral etiology.

ELIGIBILITY:
Inclusion Criteria:

* Children 1 month to 5 years old with clinical and/or radiological diagnosis of pneumonia
* Admitted to the Emergency room at the participant institutions

Exclusion Criteria:

* Prematurity
* Cardiopathy
* Pneumopathy
* Immunosuppression (congenital, chemotherapy or other cause)

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 103 (Actual)
Dates: Start 2014-01-29 (Actual); Primary Completion 2016-02-18 (Actual); Study Completion 2016-02-23 (Actual)

PRIMARY OUTCOMES:
Time of improvement of respiratory distress | From date of randomization util the date of first documented progression or date of death from any cause, whichever came first, assessed up to 10 days
  Hours since the admission to the hospital to disappear the respiratory distress
Time of improvement of oxygen desaturation | From date of randomization util the date of first documented progression or date of death from any cause, whichever came first, assessed up to 10 days
  Hours since the admission to the hospital to normalize the oxygen saturation
Time of improvement of clinical symptoms (cough, rales) | From date of randomization util the date of first documented progression or date of death from any cause, whichever came first, assessed up to 10 days
  Hours since the admission to the hospital to have improvement in clinical symptoms
Time of improvement of fever | From date of randomization util the date of first documented progression, assessed up to 10 days
  Hours to have normal temperature since the admission to the hospital
Duration of hospitalization | From date of randomization util the date of discharge or date of death from any cause, whichever came first, assessed up to 10 days
  Days for the discharge of the patient

SECONDARY OUTCOMES:
Cytokines pattern measured by flow cytometry in blood samples | From date of randomization until de date of discharge or date of death from any cause, whichever came first, assessed up to 10 days
  Th1 cytokines (interferon gamma, IL-2, tumor necrosis factor alfa) and Th2 cytokines (IL-4, IL-10, IL-6) will be determined in blood samples in 2 times: at the admission of the patient and at the discharge
Lymphoproliferation measured by incorporation of a fluorochrome in lymphocytes stimulated with Concanavalin A | From date of randomization until de date of discharge or date of death from any cause, whichever came first, assessed up to 10 days
  Blood draws will be taken at the hospital admission and at the discharge of the patient to measure the lymphoproliferative capacity of their lymphocytes by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Rosa M Wong-Chew, MD, DSc, Principal Investigator — Facultad de Medicina, Universidad Nacional Autonoma de Mexico
Locations (2):
- Mexico (2):
  - Hospital Pediatrico de Coyoacan, Mexico City, Mexico City
  - Hospital General de Mexico, México

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Acevedo-Murillo JA, Garcia Leon ML, Firo-Reyes V, Santiago-Cordova JL, Gonzalez-Rodriguez AP, Wong-Chew RM. Zinc Supplementation Promotes a Th1 Response and Improves Clinical Symptoms in Fewer Hours in Children With Pneumonia Younger Than 5 Years Old. A Randomized Controlled Clinical Trial. Front Pediatr. 2019 Nov 14;7:431. doi: 10.3389/fped.2019.00431. eCollection 2019. PMID 31803694